CLINICAL TRIAL: NCT07249619
Title: A Biopsychosocial-Based Multimodal Approach to Reducing the Risk of Delirium in Patients With Subarachnoid Hemorrhage in the Intensive Care Unit (ICU.Delibma)
Brief Title: A Biopsychosocial-Based Multimodal Approach to Reducing the Risk of Delirium in ICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emre Şenocak (Other)
Responsible Party: Sponsor-Investigator, Emre Şenocak, Assoc. Prof. Dr., Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024/6
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Subarachnoid Haemorrhagic Stroke
Keywords: Body Awareness Therapy; Communication; Delirium
MeSH Terms: conditions — Communication; Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Treatment (Active Comparator): A treatment program will be implemented in line with the recommendations of international guidelines for the treatment of delirium.
  Interventions: Other: Routine Therapy (Medical, environmental accodamation, face-to-face commucation)
- ICU.Delibma (Experimental): In addition to the treatment program implemented in line with the recommendations of international guidelines for the treatment of delirium, "Basic Body Awareness Therapy" and "Communication Program" will be applied.
  Interventions: Other: Routine Therapy (Medical, environmental accodamation, face-to-face commucation); Procedure: Biopsychosocial-Based Multimodal Approach

INTERVENTIONS:
Other: Routine Therapy (Medical, environmental accodamation, face-to-face commucation) — In the treatment of delirium, a treatment program will be implemented in line with the recommendations of international guidelines.
Procedure: Biopsychosocial-Based Multimodal Approach — Delirium treatment will be implemented in accordance with international guidelines. Additionally, a basic body awareness therapy and communication program will be implemented.
  Arms: ICU.Delibma

SUMMARY:
As part of this study, an intervention program aimed at preventing delirium in patients with subarachnoid hemorrhage treated in the intensive care unit will be implemented. Routine medical treatments, environmental adjustments, and a video-based communication program will be implemented to prevent delirium. In addition, basic body awareness training will be administered.

Patients will be divided into two groups. One group will receive only the routine treatment program recommended by international guidelines (medical, enviromental adjustment and face-to-face interview etc.), while the other group will receive body awareness therapy addition to routine interventions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-85,
* Patients scheduled for intensive care for at least 15 days due to SAH, unruptured intracranial aneurysm, and/or Arterovenous Malformation,
* Those with a Mini Mental State Examination score of > 24,
* Those with a Glasgow Coma Score of 15,
* Those with motor function in at least one extremity,
* Those with pain < 5/10 (according to the NRS)

Exclusion Criteria:

* Patients whose GCS fell to 14 or below for any reason during the study period;
* Patients who developed septic shock and MODS;
* Patients requiring endotrachial intubation and mechanical ventilation due to ARDS;
* Those requiring vasopressors such as NE at a rate of >0.25 mcg/kg/min;
* Terminal cancer cases;
* Patients with advanced chronic heart and lung failure and COPD;
* Those with a METS (exercise capacity) of <4;
* Those with a history of dementia, Alzheimer's disease, or psychiatric illness;
* Those with vision, hearing, or speech problems that would interfere with communication;
* Those with a history of epilepsy;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-01-02 (Estimated); Study Completion 2028-01-02 (Estimated)

PRIMARY OUTCOMES:
Charlson Comorbidity Index | Baseline
Charlson Comorbidity Index | 8th day after admission to ICU
Charlson Comorbidity Index | 15th day after admission to ICU
Mini-Mental State Examination Test | Baseline
APACHE II Score | Baseline
APACHE II Score | 8th day after admission to ICU
APACHE II Score | 15th day after admission to ICU
SOFA Score | Baseline
SOFA Score | 8th day after admission to ICU
SOFA Score | 15th day after admission to ICU
Glaskow Coma Score | During everyday she was admitted to the ICU
Modified Rankin Scale | Baseline
Modified Rankin Scale | 8th day after admission to ICU
Modified Rankin Scale | 15th day after admission to ICU
Simple five-item questionnaire (SARC-F) | Baseline
Simple five-item questionnaire (SARC-F) | 8th day after admission to ICU
Simple five-item questionnaire (SARC-F) | 15th day after admission to ICU
Medical Research Council Muscle Strenght | Baseline
Medical Research Council Muscle Strenght | 8th day after admission to ICU
Medical Research Council Muscle Strenght | 15th day after admission to ICU
Physical Function in Intensive Care Test (PFIT-s) | Baseline
Physical Function in Intensive Care Test (PFIT-s) | 8th day after admission to ICU
Physical Function in Intensive Care Test (PFIT-s) | 15th day after admission to ICU
Hospital Anxiety and Depression Scale | Baseline
Hospital Anxiety and Depression Scale | 8th day after admission to ICU
Hospital Anxiety and Depression Scale | 15th day after admission to ICU
Montreal Cognitive Assessment | Baseline
Montreal Cognitive Assessment | 8th day after admission to ICU
Montreal Cognitive Assessment | 15th day after admission to ICU
Nothingham Health Profile | Baseline
Nothingham Health Profile | 8th day after admission to ICU
Nothingham Health Profile | 15th day after admission to ICU
Barthel Index | Baseline
Barthel Index | 8th day after admission to ICU
Barthel Index | 15th day after admission to ICU
Modified Borg Test | During everyday she was admitted to the ICU
Confusion Assessment Method for the intensive care unit (CAM-ICU) | During everyday she was admitted to the ICU
Richmond Ajitation-Sedation Scale | During everyday she was admitted to the ICU
Numeric Rating Scale | During everyday she was admitted to the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Ulusoy, PhD, Principal Investigator — Karadeniz Technical University; Nurel Ertürk, PhD, Principal Investigator — Tarsus University; Gizem Ergün, Physiotherapist, Principal Investigator — Karadeniz Technical University; Neslihan Hatınoğlu, PhD, Principal Investigator — Karadeniz Technical University; Müge Koşucu, PhD, Principal Investigator — Karadeniz Technical University; Duygu Yıldırım, Phyiotherapist, Principal Investigator — Trabzon Kanuni Training and Research Hospital; Arzu Erden Güner, PhD, Study Chair — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Farabi Hospital, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No